CLINICAL TRIAL: NCT04054882
Title: A Randomized, Controlled, Multicenter Phase 4 Clinic Trial to Evaluate the Safety and Immunogenicity of Simultaneously Administration of sIPV and DTaP
Brief Title: Evaluation of the Safety and Immunogenicity of Simultaneously Administration of sIPV and DTaP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: China National Biotec Group Company Limited (Industry)
Collaborators: Chengdu Institute of Biological Products Co.,Ltd. (Industry); Beijing Institute of Biological Products Co Ltd. (Industry); Jiangsu Province Center for Disease Control and Prevention (Unknown); Anhui Provincial Center for Disease Control and Prevention (Unknown); Sichuan Center for Disease Control and Prevention (Other Government); Peking University (Other); National Institutes for Food and Drug Control, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: sIPV/DTaP-2019-01
Record Dates: First submitted 2019-08-09; First posted 2019-08-13 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2019-08

CONDITIONS: Vaccination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sabin-IPV and DTaP (Experimental): 234 subjects are simultaneously administrated with Sabin-IPV and DTaP at the age of 3/4/5 months old, 0.5 ml each dose, respectively
  Interventions: Biological: Sabin-IPV and DTaP
- Sabin-IPV only (Active Comparator): 234 subjects are administrated with Sabin-IPV only at the age of 3/4/5 months old, 0.5 ml each dose, respectively
  Interventions: Biological: Sabin-IPV
- DTaP only (Active Comparator): 234 subjects are administrated with DTaP only at the age of 3/4/5 months old, 0.5 ml each dose, respectively
  Interventions: Biological: DTaP

INTERVENTIONS:
Biological: Sabin-IPV and DTaP — simultaneously administration of Sabin-IPV and DTaP
  Arms: Sabin-IPV and DTaP
Biological: Sabin-IPV — administration of Sabin-IPV only
  Arms: Sabin-IPV only
Biological: DTaP — administration of DTaP only
  Arms: DTaP only

SUMMARY:
Subjects will be recruited and divided into 3 groups:(1)combined immunization of Sabin-IPV and DTaP, (2) Sabin-IPV only and (3) DTaP only.

After finishing the two basic vaccine EPI procedures, the immunogenicity and safety of both combined immunization group and individual vaccination groups will be compared and the data will be analyzed.

DETAILED DESCRIPTION:
It is recommended by China Food and Drug Administration (CFDA) that studies on simultaneous immunization of Sabin-IPV and DTaP be implemented soon and the immunogenicity and safety studies should be conducted. In China according to the current vaccination schedule, the arrangement of Sabin-IPV and DTaP falls on the same date -- at infants' 3rd and 4th months of age. In order to avoid the vaccination time conflict and explore the feasibility of simultaneous immunization, we design this phase 4 clinical trial of simultaneous vaccination of the two vaccines.

To be specific, the subjects were divided into 3 groups. Group 1 : Sabin-IPV (1st, 2nd, and 3rd doses) and DTaP (1st, 2nd, and 3rd doses) are simultaneously administrated at 3,4,5 months old ; Group 2 : subjects receive 1 dose of sIPV only at 3,4,5 months old ; Group 3 : subjects receive 1 dose of DTaP only at 3,4,5 months old .

Blood samples would be collected both before vaccination and 28-40 days after the 3rd dose of vaccination. Neutralization antibody will be detected to evaluate the seroprotection rates and antibody geometric mean concentrations. The safety of both immunization schedules will be monitored too.

ELIGIBILITY:
Inclusion Criteria:

* subjects aged 3 months old at the date of recruitment;
* with informed consent signed by parent(s) or guardians;
* parent(s) or guardians are able to attend all planned clinical appointments and
* obey and follow all study instructions;
* subjects have not been vaccinated with IPV vaccine, OPV vaccine, DTP vaccine and related vaccines;

Exclusion Criteria:

* subject who has a medical history with hypersensitiveness, eclampsia, epilepsy, cerebropathy and neurological illness;
* allergic to any ingredient of vaccine or with allergy history to any vaccine;
* subjects with immunodeficiency or suspected impairment of immunologic function (e.g. caused by HIV), or subjects are in the process of immunosuppressor therapy(Taking orally injecting of steroid hormone);
* administration of immunoglobulins within 30 days prior to this study;
* acute febrile disease(temperature ≥ 37.0°C) or infectious disease;
* have a clearly diagnosed history of thrombocytopenia or other coagulopathy,
* may cause contraindications for subcutaneous injection;
* any serious chronic illness, acute infectious diseases, or respiratory diseases;
* severe cardiovascular disease, liver and kidney diseases or diabetes mellitus with complications;
* any kind of infectious, purulent, or allergic skin diseases;
* any other factor that makes the investigator determines the subject is unsuitable for this study.

Ages: 3 Months to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 702 (Actual)
Dates: Start 2019-08-16 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2021-09-09 (Actual)

PRIMARY OUTCOMES:
Seroconversion rates at both baseline and 30 days after the 3rd vaccination | 4 months
  Determine the seroconversion rates of diphtheria, tetanus, pertussis, poliovirus (types I,II,III). Diphtheria titers are determined by toxin neutralization assay; tetanus titers are determined by enzyme-linked immunosorbent assay (ELISA)
Neutralizing antibody titers at both baseline and 30 days after the 3rd vaccination | 4 months
  Measure neutralizing antibody titers against: (1) poliovirus type I, II and III，(2) anti-pertussis toxoid ,(3) anti- FHA,(4) anti-diphtheria toxoid and (5) anti-tetanic antibodies
numbers of participants who experience adverse events | 6 months
  analyse the numbers and rates of participants who have adverse events following immunization

CONTACTS AND LOCATIONS:
Overall Officials: Fenyang Tang, Study Director — Jiangsu Provincial Center for Disease Control and Prevention
Locations (1):
- Jiangsu Provincial Center for Disease Control and Prevention, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sun X, Xu Y, Tang F, Xiao Y, Wang Z, Wang B, Zhu X, Yang X, Chen H. Immunogenicity and safety of concomitant administration of the chinese inactivated poliovirus vaccine with the diphtheria-tetanus-acellular pertussis (DTaP) vaccine in children: A multicenter, randomized, non-inferiority, controlled trial. Front Immunol. 2022 Jul 26;13:905634. doi: 10.3389/fimmu.2022.905634. eCollection 2022. PMID 35958596